CLINICAL TRIAL: NCT01362413
Title: Validation of Laboratory Test for Predicting Bone Tissue Regeneration in Patient Affected by Aseptic Pseudarthrosis and Treated With Platelet Gel
Brief Title: Validation of Laboratory Test for Predicting Bone Tissue Regeneration
Acronym: Rebone-test
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: IOR 65/10
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Nonunion of Fracture [Pseudarthrosis], Site Unspecified
Keywords: pseudarthrosis; mineralization; platelet-rich-plasma; serum
MeSH Terms: conditions — Pseudarthrosis; Calcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to determine whether the evaluation of pro-osteogenic activity of autologous serum may predict the effectiveness of platelet gel in regenerating bone tissue in patients with nonunions of long bones.

Serum samples will be collected before the surgery, and their pro-osteogenic activity will be evaluated by using a bioactivity test (mineralization assay).

In order to determine whether the pro-osteogenic activity of the serum is able to discriminate between individuals who will achieve or will not achieve bone consolidation, the laboratory results will be correlated with clinical and radiographic results at 12 months, when patients will be considered as healed or not healed.

DETAILED DESCRIPTION:
Pseudarthrosis (or 'nonunions') is defined as a bone movement which occurs after about 6 months from the traumatic event as consequence of the inadequate healing of a fracture. The use of regenerative medicine for treating recalcitrant pseudarthrosis is considered a promising strategy to promote bone consolidation. Among the various approaches used, the local cell therapy based on autologous mesenchymal stromal cells (MSC), combined with or without growth factors, has been extensively used. MSC reside within the stromal compartment of bone marrow which may be obtained from the iliac crest. Growth factors may be discharged from platelet gel (PG) which is obtained after activation of autologous platelet concentrates. Nevertheless, the results of recent clinical studies show that the above mentioned regenerative approach shows a failure rate of approximately 30% (Calori et al, 2008). The availability of a laboratory test which may predict the regenerative capacity of the PG may help the orthopaedic surgeon in addressing the decisions regarding the regenerative approach, e.g. to use or non use autologous platelet concentrates or to enhance the use of autologous derivatives with recombinant factors.The rationale for the use of platelet concentrates in pseudarthrosis is the significant reduction of osteoinductive growth factors observed at the lesion site (Gandhi et al., 2005). Platelet gel mimics what happens physiologically after any bone injury, when platelets are entrapped in a clot within a fibrin matrix. Platelet activation determines the release of various growth factors promoting bone healing. The optimal level and ratio of growth factors and their synergistic effects should be more efficient than single recombinant molecules, even though no data are available on the most relevant molecules and on their optimal amount. In this context, the in vitro mineralization assay could be a valid tool to assess the pro-osteogenic activity of platelet gel, thus obviating the measurement of the myriad of platelet-derived substances.

The aim of the study is to determine whether the evaluation of pro-osteogenic activity of autologous serum may predict the effectiveness of PG in the regeneration of bone tissue in patients with nonunions of long bones. The rationale is based on the following issues:

* in 30% of long bone nonunions treated with PG, bone consolidation is not obtained (Calori et al, 2008);
* the proportion of growth factors in serum is comparable to that observed in platelet gel after activation, even if the concentration is lower;
* the autologous serum is able to support the 'in vitro' osteogenic differentiation of MSCs and the formation of mineral nodules (mineralization assay) (Granchi et al, 2010);
* the correlation between 'in vitro' mineralization and regenerative capacity has been demonstrated in various experimental models (De Bari et al, 2008);
* preliminary data obtained in our lab showed that in patients affected by congenital pseudarthrosis of the tibia the presence of osteoinductive growth factors in serum is an essential requirement to warrant the effectiveness of the local cell therapy with MSC and PG (submitted paper).

In order to evaluate the ability of the autologous serum in inducing the mineralization in vitro the investigators will use a bioactivity test (mineralization assay). For this purpose serum samples of patients candidates to the treatment with MSC and PG will be collected the day before the surgery and used for cultivating normal MSC, whose ability to mineralize in vitro will be previously verified in standard culture conditions.

Further analysis will be conducted in order to determine whether the pro-osteogenic properties are maintained over time, and serum samples will be collected the 1 month before the surgery.

In order to determine whether the pro-osteogenic activity of the serum is able to predict and discriminate between individuals who achieve or not achieve bone consolidation, the laboratory results will be correlated with clinical and radiographic results at 12 months, when patients will be considered as healed or not healed.

ELIGIBILITY:
Eligible patients will be identified according to the following criteria.

Inclusion criteria:

* patients with aseptic nonunion of long bones and candidates for treatment with platelet gel and MSC in addition to fixation devices and bone grafting;
* patients who have given their written consent to participate in the study.

Exclusion criteria:

* patients with bone infections;
* patients with congenital disorders involving the skeletal development;
* patients treated with corticosteroids or other immunosuppressive agents;
* patients suffering from mental or psychiatric disorders that preclude the possibility of correctly adhering to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Correlation between laboratory results at the surgery and clinical and radiographic results at 12 months, when patients will be considered as healed or not healed. | 13 months, for each patient
  The pro-osteogenic ability of autologous serum will be evaluated by using a bioactivity test (mineralization assay). For this purpose serum samples will be collected 1 day before the surgery and used for culturing osteogenic cells. The ability of inducing the mineralization will be assessed after 10 days of culture.
  At 12 months, clinical outcome will be evaluated as follows:
  * anteroposterior and lateral X-rays to assess the continuity of bone in the various plans;
  * semeiotics of the consolidation;
  * assessment of pain during loading (Visual Analogue Scale).

SECONDARY OUTCOMES:
Assessment of the pro-osteogenic properties of serum over time. | 1 month before surgery
  In order to determine whether the pro-osteogenic properties are maintained over time, we planned to collect other serum samples, namely preoperatively, 1 month before the surgery.
  The pro-osteogenic activity will be evaluated as previously described.
Correlation between laboratory testing and timing of healing. | 1, 3, 6, and 9 months postoperatively
  Clinical and radiographic results will be assessed at intermediate end points, as previously described.

CONTACTS AND LOCATIONS:
Overall Officials: Donatella Granchi, MD, Principal Investigator — Laboratorio di Fisiopatologia Ortopedica e Medicina Rigenerativa - Istituto Ortopedico Rizzoli; Dante Dallari, MD, Principal Investigator — Centro di Riferimento Specialistico di Applicazioni Cliniche di Medicina Rigenerativa in Ortopedia - Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

REFERENCES:
- [Background] Gandhi A, Bibbo C, Pinzur M, Lin SS. The role of platelet-rich plasma in foot and ankle surgery. Foot Ankle Clin. 2005 Dec;10(4):621-37, viii. doi: 10.1016/j.fcl.2005.06.009. PMID 16297823
- [Background] Calori GM, Tagliabue L, Gala L, d'Imporzano M, Peretti G, Albisetti W. Application of rhBMP-7 and platelet-rich plasma in the treatment of long bone non-unions: a prospective randomised clinical study on 120 patients. Injury. 2008 Dec;39(12):1391-402. doi: 10.1016/j.injury.2008.08.011. Epub 2008 Nov 22. PMID 19027898
- [Background] Cenni E, Savarino L, Perut F, Fotia C, Avnet S, Sabbioni G. Background and rationale of platelet gel in orthopaedic surgery. Musculoskelet Surg. 2010 May;94(1):1-8. doi: 10.1007/s12306-009-0048-9. Epub 2009 Nov 24. PMID 19937168
- [Background] Arvidson K, Abdallah BM, Applegate LA, Baldini N, Cenni E, Gomez-Barrena E, Granchi D, Kassem M, Konttinen YT, Mustafa K, Pioletti DP, Sillat T, Finne-Wistrand A. Bone regeneration and stem cells. J Cell Mol Med. 2011 Apr;15(4):718-46. doi: 10.1111/j.1582-4934.2010.01224.x. PMID 21129153
- [Background] De Bari C, Dell'Accio F, Karystinou A, Guillot PV, Fisk NM, Jones EA, McGonagle D, Khan IM, Archer CW, Mitsiadis TA, Donaldson AN, Luyten FP, Pitzalis C. A biomarker-based mathematical model to predict bone-forming potency of human synovial and periosteal mesenchymal stem cells. Arthritis Rheum. 2008 Jan;58(1):240-50. doi: 10.1002/art.23143. PMID 18163504
- [Background] Granchi D, Devescovi V, Baglio SR, Leonardi E, Donzelli O, Magnani M, Stilli S, Giunti A, Baldini N. Biological basis for the use of autologous bone marrow stromal cells in the treatment of congenital pseudarthrosis of the tibia. Bone. 2010 Mar;46(3):780-8. doi: 10.1016/j.bone.2009.10.044. Epub 2009 Nov 10. PMID 19900596
- See also: Istituto Ortopedico Rizzoli - Home Page — http://www.ior.it/